CLINICAL TRIAL: NCT02831413
Title: Testing the Effectiveness of Relationship Smarts Curriculum and the Effects of Enhanced Facilitator Training
Brief Title: Testing the Effectiveness of Relationship Smarts and the Effects of Enhanced Facilitator Training
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPR-500098-FB
Record Dates: First submitted 2016-06-02; First posted 2016-07-13 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Knowledge; Attitude
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): Control group members will receive an alternate curriculum that is not related to relationship education. Family Bridges has identified a computer programming curriculum, Codeacademy, that teaches students how to use HTML.
  Interventions: Behavioral: Codeacademy
- RS+ (Experimental): The RS+ curriculum's 12 sessions will be delivered over a period of about 12 weeks during the winter quarter, with an average of one session taught per week. The lessons cover topics such as personal values, the principals of smart relationships, communication and conflict management, and sexual decision making.
  Interventions: Behavioral: RS+
- RS+ with enhanced facilitator support (Experimental): The RS+ curriculum's 12 sessions will be delivered over a period of about 12 weeks during the winter quarter, with an average of one session taught per week. The lessons cover topics such as personal values, the principals of smart relationships, communication and conflict management, and sexual decision making. Affiliates assigned to this enhanced treatment group will participate in enhanced facilitator training and support activities.
  Interventions: Behavioral: RS+

INTERVENTIONS:
Behavioral: RS+ — The curriculum's 12 sessions will be delivered over a period of about 12 weeks during the winter quarter, with an average of one session taught per week. The lessons cover topics such as personal values, the principals of smart relationships, communication and conflict management, and sexual decision making.
  Arms: RS+; RS+ with enhanced facilitator support
Behavioral: Codeacademy — a computer programming curriculum, Codeacademy, that teaches students how to use HTML.
  Arms: Control

SUMMARY:
This project will test the effectiveness of offering healthy marriage and relation education for youth as part of the regular school curriculum and examine whether providing enhanced training and support for facilitators shows promise for enhancing the effects on high school students. The evaluation will examine a range of students' relationship outcomes, including their attitudes toward relationships, their knowledge of healthy relationships, their communication skills, and the characteristics of their current relationship.

DETAILED DESCRIPTION:
Family Bridges will deliver the "Relationship Smarts +" program to students at 10 Chicago-area high schools. The RS+ curriculum will be delivered to 9th grade students in the target schools and classrooms during the 2016-2017 and 2017-2018 school years. The curriculum's 12 sessions will be delivered over a period of about 12 weeks during the winter quarter, with an average of one session taught per week.The lessons cover topics such as personal values, the principals of smart relationships, communication and conflict management, and sexual decision making. Using a three-arm randomized controlled trial design, this study will test the effectiveness of offering RS+ as part of the regular school curriculum on the students' knowledge of healthy relationships, their communication skills, and the characteristics of their current relationship. In addition to testing the effects of the curriculum, the study will also test the effects of providing enhanced training and support to facilitators.

ELIGIBILITY:
Inclusion Criteria:

* Students must be age 17 or younger
* have consent from a parent or guardian for evaluation activities
* provide assent for evaluation activities.

Exclusion Criteria:

* Students in evaluation classrooms who do not meet these criteria will still receive programming, but will not be included in the STREAMS data collection activities or in the study's analysis.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Knowledge about Healthy Relationships | end of programming (approx. 12 weeks after beginning of programming )
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.
Attitudes about Healthy Relationships | end of programming (approx. 12 weeks after beginning of programming )
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.
Knowledge about Healthy Relationships | 1 year follow-up
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.
Attitudes about Healthy Relationships | 1 year follow-up
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.

SECONDARY OUTCOMES:
Communications skills | end of programming (approx. 12 weeks after beginning of programming )
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.
Characteristics of current romantic relationship | end of programming (approx. 12 weeks after beginning of programming )
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.
Communications skills | 1 year follow-up
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.
Characteristics of current romantic relationship | 1 year follow-up
  audio computer-assisted self-administered interviewing (ACASI) software on tablet devices.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Paulsell, Principal Investigator — Mathematica Policy Research
Locations (1):
- Family Bridges, Inc., Oak Park, Illinois, United States

IPD SHARING:
Plan to Share IPD: No